CLINICAL TRIAL: NCT02119715
Title: A Phase II Study Comparing Pegylated rhG-CSF（HHPG-19K） and rhG-CSF as Supportive Therapy to Breast Cancer Patients Receiving Neoadjuvant/Adjuvant Chemotherapy
Brief Title: A Phase II Study Comparing Pegylated rhG-CSF（HHPG-19K） and rhG-CSF in Breast Cancer Patients Receiving Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HHPG-19K-II-01
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Breast Cancer; Neutropenia; Febrile Neutropenia
Keywords: Breast Cancer; Neutropenia; Febrile Neutropenia
MeSH Terms: conditions — Breast Neoplasms; Neutropenia; Febrile Neutropenia | interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pegylated rhG-CSF 100μg/kg (Experimental): Chemotherapy naive patients receiving chemotherapy and Pegylated rhG-CSF（HHPG-19K） 100µg/kg in cycle 2 to 4
  Interventions: Drug: Pegylated rhG-CSF 100μg/kg
- Pegylated rhG-CSF 150μg/kg (Experimental): Chemotherapy naive patients receiving chemotherapy and Pegylated rhG-CSF（HHPG-19K)150 μg/kg in cycle 2 to 4
  Interventions: Drug: Pegylated rhG-CSF:150 μg/kg
- G-CSF 5 μg/kg/d (Active Comparator): Chemotherapy naive patients receiving chemotherapy and rhG-CSF 5μg/kg/day in cycle 2 to 4
  Interventions: Drug: rhG-CSF 5 μg/kg/day

INTERVENTIONS:
Drug: Pegylated rhG-CSF 100μg/kg — Patients were administered pegylated rhG-CSF 100 ug/kg once at the 3rd day of 2 to 4 chemotherapy cycle(epirubicin 75mg/m2+docetaxel 75mg/m2 for neoadjuvant therapy and epirubicin 100mg/m2+cyclophosphamide 600mg/m2 for adjuvant therapy).
  Other Names: HHPG-19K 100µg/kg
  Arms: Pegylated rhG-CSF 100μg/kg
Drug: Pegylated rhG-CSF:150 μg/kg — Patients were administered pegylated rhG-CSF 150 ug/kg once at the 3rd day of 2 to 4 chemotherapy cycle(epirubicin 75mg/m2+docetaxel 75mg/m2 for neoadjuvant therapy and epirubicin 100mg/m2+cyclophosphamide 600mg/m2 for adjuvant therapy).
  Other Names: HHPG-19K 150μg/kg
  Arms: Pegylated rhG-CSF 150μg/kg
Drug: rhG-CSF 5 μg/kg/day — Patients were administered rhG-CSF 5 ug/kg daily during chemotherapy cycle(epirubicin 75mg/m2+docetaxel 75mg/m2 for neoadjuvant therapy and epirubicin 100mg/m2+cyclophosphamide 600mg/m2 for adjuvant therapy) until (1)continuous injection for 14 days (2)two successive ANC counts exceed 5.0×109/L（3）ANC counts exceed 15×109/L at anytime.
  Other Names: Jie Xin 5 μg/kg/day
  Arms: G-CSF 5 μg/kg/d

SUMMARY:
Neutropenia is one of the most frequent adverse effects of chemotherapy, and the main factor to limit the dosage and the continuation of chemotherapy. A newly pegylated rhG-CSF was independently developed by JIANGSU HENGRUI Medicine Co., Ltd, China. Phase 1a, 1b trials have shown that pegylated rhG-CSF has decreased renal clearance, increased plasma half-life, and prolonged efficacy in compare with rhG-CSF. The purpose of this study is to determine the safety and effectiveness of pegylated rhG-CSF in preventing neutropenia following chemotherapy in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathology diagnosis of breast cancer,Chemotherapy naïve
* ECOG performance status 0-1
* Age 18 to 70 years
* Available for at least 2 cycles of consistent neoadjuvant/adjuvant therapy
* White blood cell ≥ 4.0×109/L; absolute neutrophil count ≥2.0 × 109/L; platelet count ≥ 100 × 109/L
* Alanine aminotransferase ≤1.5×ULN; aspartate aminotransferase ≤1.5×ULN; serum creatinine ≤1.5×ULN
* No obvious cardiac dysfunction

Exclusion Criteria:

* Prior bone marrow or stem cell transplantation
* Received systemic antibiotics treatment within 72 h of chemotherapy
* Other disease might have influence on bone marrow function
* Radiation therapy within 4 weeks of randomization into this study
* Previous exposure or or allergic to Pegylated rhG-CSF
* Pregnancy, lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Incidence and the duration of grade 3/4 neutropenia in cycle 2 and the time frame of ANC recovery to 2.0×109/L | 6 weeks
  Proportion and the duration of subjects developing ANC lower than 1.0×109/L

SECONDARY OUTCOMES:
Incidence of the febrile neutropenia in cycle 1 and cycle 2 | 6 weeks
  Rate of ANC<0.5×109/L and auxiliary temperature>38.5℃
ANC alteration in cycle 1 and cycle 2 | 6 weeks
  Weekly laboratory ANC value alteration

CONTACTS AND LOCATIONS:
Overall Officials: ZeFei Jiang, M.D, Principal Investigator — 307 Hospital Affiliated to Academy Military Medical Science
Locations (1):
- 307 Hospital Affiliated to Academy Military Medical Science, Beijing, China